CLINICAL TRIAL: NCT02354170
Title: Short-Term Oral Mifepristone for Central Serous Chorioretinopathy. A Placebo-controlled Dose Ranging Study of Mifepristone in the Treatment of CSC (STOMP-CSC)
Brief Title: Short-Term Oral Mifepristone for Central Serous Chorioretinopathy
Acronym: STOMP-CSC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roger Goldberg, M.D., MBA (Other)
Collaborators: Ophthalmic Consultants of Boston (Other)
Responsible Party: Sponsor-Investigator, Roger Goldberg, M.D., MBA, Ophthalmologist, Retina and Vitreous, Bay Area Retina Associates
Organization: Bay Area Retina Associates (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: STOMP-CSC
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Central Serous Chorioretinopathy
Keywords: Central Serous Chorioretinopathy, CSC
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (m300) (Experimental): One (1) 300-mg mifepristone tablet, taken once daily for 4 weeks
  Interventions: Drug: Mifepristone
- Cohort 2 (m900) (Experimental): Three (3) 300-mg mifepristone tablets (900-mg dose), taken once daily for 4 weeks
  Interventions: Drug: Mifepristone
- Cohort 3 (Placebo) (Placebo Comparator): Placebo taken once daily for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mifepristone
  Arms: Cohort 1 (m300); Cohort 2 (m900)
Drug: Placebo
  Arms: Cohort 3 (Placebo)

SUMMARY:
The goal of the study is to assess the efficacy and safety of mifepristone 300 or 900-mg once-daily dosing by mouth for 4 weeks in patients with central serous chorioretinopathy.

DETAILED DESCRIPTION:
* Prospective, randomized, double-masked, placebo-controlled dose-ranging study
* Eligible patients will be those with CSC, with symptoms of blurred or distorted vision, with the presence of sub-retinal fluid as documented on optical coherence tomography (OCT) in the central foveal sub-field
* Only one eye of a participant will be included in the study, although both eyes will be evaluated. In patients with bilateral CSC, the eye with more sub-foveal fluid on OCT will be the study eye.
* Patients will be evaluated and treated at one of two study centers:

Ophthalmic Consultants of Boston (OCB), 50 Staniford St., Suite 600, Boston, MA

Bay Area Retina Associates (BARA), 122 La Casa Via, Suite 223, Walnut Creek, CA

* All participants will receive a standard ophthalmic examination as well as fluorescein and indocyanine green angiography and macular OCT per protocol.
* 30 patients will be enrolled, as follows:

  10 patients will be randomly assigned to Cohort 1, and will take one (1) mifepristone 300-mg tablet (300 mg total dose) once daily by mouth for 4 weeks.

  10 patients will be randomly assigned to Cohort 2, and will take three (3) mifepristone 300-mg tablet (900 mg total dose) once daily by mouth for 4 weeks.

  10 patients will be randomly assigned to Cohort 3, and will take placebo tablet(s) once daily by mouth for 4 weeks.
* After completing the enrollment criteria, a subject will be randomized 1:1:1 to Cohort 1, 2, or 3.
* During the Baseline visit and at the Week 2, 4, and 8 visits, all subjects will have laboratory testing of the following lab tests: serum electrolytes, BUN and creatinine, liver function tests
* Prior to initiating dosing of the study drug, all women of child-bearing potential (WOCBP) will have a serum beta-HCG assessed to rule out pregnancy; all WOCBP who are enrolled in the study will be required to use barrier contraception throughout the study.
* Adverse events will be tracked at each visit (see "Data Safety and Monitoring Plan" below)

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of central serous chorioretinopathy (CSC) with symptoms 6 weeks or prior documented episodes of sub-retinal fluid; patients who have had previous treatment for CSC may be included
2. Presence of sub-retinal fluid as documented on optical coherence tomography (OCT) in the central foveal sub-field
3. Age 18 or over
4. Willing and able to comply with clinic visits and study-related procedures
5. Ability to give written informed consent

Exclusion Criteria:

1. Age less than 18
2. Persons with impaired decision-making ability.
3. Women who are known to be breast-feeding, pregnant or are actively trying to conceive.
4. Additional eye disease affecting the macula, posterior retina, or ocular media that would limit or prevent the acquisition of OCT and angiographic images.
5. At screening, serum potassium < LLN, BUN > 1.5 ULN, serum creatinine >1.5 ULN, AST > 1.5 ULN, ALT >1.5 ULN, bilirubin > 1.5 ULN, alkaline phosphatase > 1.5 ULN, serum albumin >1.5 ULN or <LLN.
6. Intraocular surgery (including cataract surgery) in the study eye within 60 days preceding baseline.
7. Active intraocular inflammation (grade trace or above) in the study eye.
8. Patients taking simvastatin, lovastatin, and CYP3A substrates with narrow therapeutic ranges, such as cyclosporine, dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus, and tacrolimus.
9. Patients who require concomitant treatment with systemic corticosteroids for serious medical conditions or illnesses (e.g., immunosuppression after organ transplantation).
10. Women with a history of unexplained vaginal bleeding and women with endometrial hyperplasia with atypia or endometrial carcinoma.
11. Patients with prior hypersensitivity reactions to mifepristone or to any of the product components.
12. Patients with known hypersensitivity to fluorescein or indocyanine green dyes.

    * WOCBP must be willing to practice adequate contraception during the study (adequate contraceptive measures include intrauterine device [IUD]; bilateral tubal ligation; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly). Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Resolution of Sub-retinal Fluid | 4 weeks after treatment
  Presence or absence of subretinal fluid on spectral-domain OCT after 4 weeks of treatment with mifepristone 300 or 900 mg daily, compared with placebo.

SECONDARY OUTCOMES:
Change in sub-retinal fluid and/or intraretinal fluid | Week 1, 2, 4, and 8
  Change compared to Baseline in subretinal fluid and/or intraretinal fluid on OCT at Week 1, 2, 4, and 8,
Best Corrected Visual Acuity | Week 1, 2, 4, and 8
  Change compared to Baseline in ETDRS BCVA at Week 1, 2, 4, and 8.
Change in macular thickness | Week 1, 2, 4, and 8
  Change compared to Baseline in central macular circle thickness on OCT, automatically calculated with OCT software at Week 1, 2, 4, and 8.
Change in foveal thickness | Week 1, 2, 4, and 8
  Change compared to Baseline in thickness of subretinal fluid under the fovea on OCT, manually calculated at Week 1, 2, 4, and 8
Change in choroidal thickness | Week 1, 2, 4, and 8
  Change compared to Baseline in thickness of choroid under the fovea on enhanced-depth imaging OCT, manually calculated, at Week 1, 2, 4, and 8.
Dye leakage in vasculature | Week 4 and 8
  Change compared to Baseline in dye leakage characteristics on fluorescein and indocyanine green angiography at Week 4 and Week 8.
Change in OCT characteristics in the fellow eye | Week 8
  Change compared to Baseline in the same OCT characteristics listed above, in the fellow eye.
Proportion of acute vs. chronic CSC patients | Week 8
  Proportion of acute versus chronic CSC patients as determined at Baseline, with the above outcomes analyzed for each sub-group.
Safety and Tolerability Characteristics | Week 8
  Safety and tolerability characteristics in this patient population via clinical laboratory data and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Roger A Goldberg, M.D., MBA, Principal Investigator — Bay Area Retina Associates; Jeffrey S Heier, M.D., Principal Investigator — Ophthalmic Consultants of Boston
Locations (2):
- United States (2):
  - Bay Area Retina Associates, Walnut Creek, California
  - Ophthalmic Consultants of Boston, Boston, Massachusetts

REFERENCES:
- [Background] Zhao M, Celerier I, Bousquet E, Jeanny JC, Jonet L, Savoldelli M, Offret O, Curan A, Farman N, Jaisser F, Behar-Cohen F. Mineralocorticoid receptor is involved in rat and human ocular chorioretinopathy. J Clin Invest. 2012 Jul;122(7):2672-9. doi: 10.1172/JCI61427. Epub 2012 Jun 11. PMID 22684104
- [Background] Gemenetzi M, De Salvo G, Lotery AJ. Central serous chorioretinopathy: an update on pathogenesis and treatment. Eye (Lond). 2010 Dec;24(12):1743-56. doi: 10.1038/eye.2010.130. Epub 2010 Oct 8. PMID 20930852
- [Background] Bouzas EA, Karadimas P, Pournaras CJ. Central serous chorioretinopathy and glucocorticoids. Surv Ophthalmol. 2002 Sep-Oct;47(5):431-48. doi: 10.1016/s0039-6257(02)00338-7. PMID 12431693
- [Background] Tittl MK, Spaide RF, Wong D, Pilotto E, Yannuzzi LA, Fisher YL, Freund B, Guyer DR, Slakter JS, Sorenson JA. Systemic findings associated with central serous chorioretinopathy. Am J Ophthalmol. 1999 Jul;128(1):63-8. doi: 10.1016/s0002-9394(99)00075-6. PMID 10482095
- [Background] Yannuzzi LA. Type-A behavior and central serous chorioretinopathy. Retina. 1987 Summer;7(2):111-31. doi: 10.1097/00006982-198700720-00009. PMID 3306853
- [Background] Spaide RF, Campeas L, Haas A, Yannuzzi LA, Fisher YL, Guyer DR, Slakter JS, Sorenson JA, Orlock DA. Central serous chorioretinopathy in younger and older adults. Ophthalmology. 1996 Dec;103(12):2070-9; discussion 2079-80. doi: 10.1016/s0161-6420(96)30386-2. PMID 9003341
- [Background] Ross A, Ross AH, Mohamed Q. Review and update of central serous chorioretinopathy. Curr Opin Ophthalmol. 2011 May;22(3):166-73. doi: 10.1097/ICU.0b013e3283459826. PMID 21427570
- [Background] Castro-Correia J, Coutinho MF, Rosas V, Maia J. Long-term follow-up of central serous retinopathy in 150 patients. Doc Ophthalmol. 1992;81(4):379-86. doi: 10.1007/BF00169099. PMID 1486812
- [Background] Gilbert CM, Owens SL, Smith PD, Fine SL. Long-term follow-up of central serous chorioretinopathy. Br J Ophthalmol. 1984 Nov;68(11):815-20. doi: 10.1136/bjo.68.11.815. PMID 6541945
- [Background] Bujarborua D. Long-term follow-up of idiopathic central serous chorioretinopathy without laser. Acta Ophthalmol Scand. 2001 Aug;79(4):417-21. doi: 10.1034/j.1600-0420.2001.079004417.x. PMID 11453866
- [Background] Folk JC, Thompson HS, Han DP, Brown CK. Visual function abnormalities in central serous retinopathy. Arch Ophthalmol. 1984 Sep;102(9):1299-302. doi: 10.1001/archopht.1984.01040031049021. PMID 6477246
- [Background] Chan WM, Lai TY, Lai RY, Liu DT, Lam DS. Half-dose verteporfin photodynamic therapy for acute central serous chorioretinopathy: one-year results of a randomized controlled trial. Ophthalmology. 2008 Oct;115(10):1756-65. doi: 10.1016/j.ophtha.2008.04.014. Epub 2008 Jun 5. PMID 18538401
- [Background] Spitznas M, Huke J. Number, shape, and topography of leakage points in acute type I central serous retinopathy. Graefes Arch Clin Exp Ophthalmol. 1987;225(6):437-40. doi: 10.1007/BF02334172. PMID 3678855
- [Background] Fujimoto H, Gomi F, Wakabayashi T, Sawa M, Tsujikawa M, Tano Y. Morphologic changes in acute central serous chorioretinopathy evaluated by fourier-domain optical coherence tomography. Ophthalmology. 2008 Sep;115(9):1494-500, 1500.e1-2. doi: 10.1016/j.ophtha.2008.01.021. Epub 2008 Apr 18. PMID 18394706
- [Background] Montero JA, Ruiz-Moreno JM. Optical coherence tomography characterisation of idiopathic central serous chorioretinopathy. Br J Ophthalmol. 2005 May;89(5):562-4. doi: 10.1136/bjo.2004.049403. PMID 15834085
- [Background] Imamura Y, Fujiwara T, Margolis R, Spaide RF. Enhanced depth imaging optical coherence tomography of the choroid in central serous chorioretinopathy. Retina. 2009 Nov-Dec;29(10):1469-73. doi: 10.1097/IAE.0b013e3181be0a83. PMID 19898183
- [Background] Robertson DM, Ilstrup D. Direct, indirect, and sham laser photocoagulation in the management of central serous chorioretinopathy. Am J Ophthalmol. 1983 Apr;95(4):457-66. doi: 10.1016/0002-9394(83)90265-9. PMID 6682293
- [Background] Ficker L, Vafidis G, While A, Leaver P. Long-term follow-up of a prospective trial of argon laser photocoagulation in the treatment of central serous retinopathy. Br J Ophthalmol. 1988 Nov;72(11):829-34. doi: 10.1136/bjo.72.11.829. PMID 3061449
- [Background] Taban M, Boyer DS, Thomas EL, Taban M. Chronic central serous chorioretinopathy: photodynamic therapy. Am J Ophthalmol. 2004 Jun;137(6):1073-80. doi: 10.1016/j.ajo.2004.01.043. PMID 15183792
- [Background] Inoue R, Sawa M, Tsujikawa M, Gomi F. Association between the efficacy of photodynamic therapy and indocyanine green angiography findings for central serous chorioretinopathy. Am J Ophthalmol. 2010 Mar;149(3):441-6.e1-2. doi: 10.1016/j.ajo.2009.10.011. PMID 20172070
- [Background] Maruko I, Iida T, Sugano Y, Ojima A, Ogasawara M, Spaide RF. Subfoveal choroidal thickness after treatment of central serous chorioretinopathy. Ophthalmology. 2010 Sep;117(9):1792-9. doi: 10.1016/j.ophtha.2010.01.023. Epub 2010 May 15. PMID 20472289
- [Background] Reibaldi M, Cardascia N, Longo A, Furino C, Avitabile T, Faro S, Sanfilippo M, Russo A, Uva MG, Munno F, Cannemi V, Zagari M, Boscia F. Standard-fluence versus low-fluence photodynamic therapy in chronic central serous chorioretinopathy: a nonrandomized clinical trial. Am J Ophthalmol. 2010 Feb;149(2):307-315.e2. doi: 10.1016/j.ajo.2009.08.026. Epub 2009 Nov 6. PMID 19896635
- [Background] Shin JY, Woo SJ, Yu HG, Park KH. Comparison of efficacy and safety between half-fluence and full-fluence photodynamic therapy for chronic central serous chorioretinopathy. Retina. 2011 Jan;31(1):119-26. doi: 10.1097/IAE.0b013e3181e378f2. PMID 20890242
- [Background] Golshahi A, Klingmuller D, Holz FG, Eter N. Ketoconazole in the treatment of central serous chorioretinopathy: a pilot study. Acta Ophthalmol. 2010 Aug;88(5):576-81. doi: 10.1111/j.1755-3768.2008.01467.x. Epub 2009 May 12. PMID 19456313
- [Background] Nielsen JS, Jampol LM. Oral mifepristone for chronic central serous chorioretinopathy. Retina. 2011 Oct;31(9):1928-36. doi: 10.1097/IAE.0b013e31821c3ef6. PMID 21878843
- [Background] Forooghian F, Meleth AD, Cukras C, Chew EY, Wong WT, Meyerle CB. Finasteride for chronic central serous chorioretinopathy. Retina. 2011 Apr;31(4):766-71. doi: 10.1097/IAE.0b013e3181f04a35. PMID 21273946
- [Background] Avci R, Deutman AF. [Treatment of central serous choroidopathy with the beta receptor blocker metoprolol (preliminary results)]. Klin Monbl Augenheilkd. 1993 Mar;202(3):199-205. doi: 10.1055/s-2008-1045583. German. PMID 8510413
- [Background] Tatham A, Macfarlane A. The use of propranolol to treat central serous chorioretinopathy: an evaluation by serial OCT. J Ocul Pharmacol Ther. 2006 Apr;22(2):145-9. doi: 10.1089/jop.2006.22.145. PMID 16722801
- [Background] Pikkel J, Beiran I, Ophir A, Miller B. Acetazolamide for central serous retinopathy. Ophthalmology. 2002 Sep;109(9):1723-5. doi: 10.1016/s0161-6420(02)01157-0. PMID 12208723
- [Background] Davis KL, Nappi JM. The cardiovascular effects of eplerenone, a selective aldosterone-receptor antagonist. Clin Ther. 2003 Nov;25(11):2647-68. doi: 10.1016/s0149-2918(03)80326-0. PMID 14693297
- [Background] McCurley A, Jaffe IZ. Mineralocorticoid receptors in vascular function and disease. Mol Cell Endocrinol. 2012 Mar 24;350(2):256-65. doi: 10.1016/j.mce.2011.06.014. Epub 2011 Jun 24. PMID 21723914
- [Background] Pitt B, Remme W, Zannad F, Neaton J, Martinez F, Roniker B, Bittman R, Hurley S, Kleiman J, Gatlin M; Eplerenone Post-Acute Myocardial Infarction Heart Failure Efficacy and Survival Study Investigators. Eplerenone, a selective aldosterone blocker, in patients with left ventricular dysfunction after myocardial infarction. N Engl J Med. 2003 Apr 3;348(14):1309-21. doi: 10.1056/NEJMoa030207. Epub 2003 Mar 31. PMID 12668699
- [Background] Weinberger MH, Roniker B, Krause SL, Weiss RJ. Eplerenone, a selective aldosterone blocker, in mild-to-moderate hypertension. Am J Hypertens. 2002 Aug;15(8):709-16. doi: 10.1016/s0895-7061(02)02957-6. PMID 12160194
- [Background] Krum H, Nolly H, Workman D, He W, Roniker B, Krause S, Fakouhi K. Efficacy of eplerenone added to renin-angiotensin blockade in hypertensive patients. Hypertension. 2002 Aug;40(2):117-23. doi: 10.1161/01.hyp.0000025146.19104.fe. PMID 12154100
- [Background] Flack JM, Oparil S, Pratt JH, Roniker B, Garthwaite S, Kleiman JH, Yang Y, Krause SL, Workman D, Saunders E. Efficacy and tolerability of eplerenone and losartan in hypertensive black and white patients. J Am Coll Cardiol. 2003 Apr 2;41(7):1148-55. doi: 10.1016/s0735-1097(03)00054-8. PMID 12679215
- [Derived] Lange CA, Qureshi R, Pauleikhoff L. Interventions for central serous chorioretinopathy: a network meta-analysis. Cochrane Database Syst Rev. 2025 Jun 16;6(6):CD011841. doi: 10.1002/14651858.CD011841.pub3. PMID 40522203